CLINICAL TRIAL: NCT04835779
Title: Biometric and Biological Data for Diagnosis and Therapy of Pain Patients German: Biometrische Und Biologische Daten für Die Diagnose Und Therapie Bei Schmerzpatienten
Brief Title: Biometric and Biological Data for Diagnosis and Therapy of Pain Patients
Acronym: Bio2Treat
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Roman Rolke, Direktor Klinik für Palliativmedizin, RWTH Aachen University
Other Study IDs: 18-018
Record Dates: First submitted 2021-02-11; First posted 2021-04-08 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Small Fiber Neuropathy
Keywords: Pain; SFN
MeSH Terms: conditions — Small Fiber Neuropathy; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- SFN Patients: Patients with diagnosed Small Fibre Neuropathy
- Patients undergoing chemotherapy: Patients undergoing chemotherapy and are expected to develop SFN as a result
- Healthy Volunteer: Healthy test person
- Healthy Volunteer PREPs: For the pain-evoked potentials (PREPs), 20 additional healthy control subjects are to be included. Four subjects (2 male, 2 female) from each of the age decades 20-29, 30-39, 40-49, 50-59, 60-69.

SUMMARY:
In order to meet the challenge of an unambiguous diagnosis and effective therapy of SFN or the prognosis of susceptibility to the development of SFN, this project aims to create a data basis on which software will be developed during the project. This software should later be able to combine (integrate) quantifiable biometric data collected from the patient (both objectively measured and patient reported parameters) with the results of biological analyses of the patient's own nerve cells from stem cells. We expect that the patient-specific combination and correlation of biometric and biological data can lead to a significant improvement in the diagnosis, prognosis and therapy of chronic pain. The initial data collection required for the development of such a software (Bio2Integrate) will be carried out in three different project parts: Bio2Watch, Bio2Patient and Bio2Cell

DETAILED DESCRIPTION:
Bio2Watch: In this clinical project part biometric patient data of 24 SFN patients, 3 cancer patients and 21 subjects (control group) will be collected for a period of one year using a PainWatch. The term PainWatch includes an Apple Watch 5 with iPhone 8 and installed app for pain recording. With the aid of the PainWatch, the personal pain sensation in everyday life is documented and personal data such as the pulse rate and the daily number of steps, as well as environmental data, such as the prevailing air pressure, humidity and temperature are recorded. The aim is to use these data as a basis for initial indications of pain-inducing stimuli or combinations of stimuli.

Bio2Patient: In this clinical project part clinically quantifiable tests are carried out, such as quantitative sensory testing (QST), which examines subjective thermal and mechanical sensory perception and pain thresholds. The goal is to determine a specific pain phenotype. In addition, pain evoked potentials (PREPs) are performed to draw conclusions about the function of thin nerve fibers (pain fibers), including projection to the brain. Supplementary SF-36 pain questionnaires are completed to assess the quality of life.For the pain-evoked potentials (PREPs), a total of 20 additional healthy control subjects are to be included (control group D). Four subjects (2 male, 2 female) from each of the age decades 20-29, 30-39, 40-49, 50-59, 60-69 will be included.

Bio2Cell: In the cell-based project part induced pluripotent stem cells (iPS cells) are produced from blood cells of SFN patients, cancer patients and volunteers. These cells will be differentiated into sensory neurons that are relevant in pain processing, so-called nociceptors. Since these nociceptors are derived from the individual patient, they carry the individual genetic characteristics of the patient. These neurons are then analyzed by multi-electrode arrays (MEA). With this method environmental influences such as temperature and air pressure or drugs on the pathophysiology of the patient's are investigated. The main goal is to simulate the conditions, which lead to pain sensation in the context of Bio2Watch and Bio2Patient.

Bio2Integrate: The results from Bio2Watch, Bio2Patient and Bio2Cell will then flow into the software to be developed during the project. Thus, in addition to the identification of stimuli that stimulate pain as well as a genetic correlation to certain markers will be possible. In addition, the targeted modification of the cellular properties of the patient's own sensory neurons through the application of the chemotherapeutic agent can be investigated. To this end, measurements will be made on the cells before and after the application of the substance and compare them with each other. This is the basis for components of the "machine learning " of the Bio2Integrate software.The results of the clinical subprojects are thus an essential component of Bio2Integrate.

ELIGIBILITY:
Inclusion Criteria:

Group A: Criteria 1-5 Group B: Criteria 2-5 Group C: Criteria 2-6 Group D: Criteria 2-4

1. Small fiber neuropathy (after clinical examination or QST or skin biopsy findings)
2. Legal age
3. Written declaration of consent
4. Persons who are legally competent and mentally capable of following the instructions of the staff
5. Sufficient affinity for independent handling of the technology used (PainWatch incl. the corresponding apps) for daily digital pain recording
6. Imminent initiation of neurotoxic chemotherapy in cancer with solid tumors (preferably of the gastrointestinal tract) There are no plans for follow-up recruitment in case no neuropathy develops after chemo.

Exclusion Criteria:

For all Groups:

1. Persons who are accommodated in an institution by order of the authorities or courts
2. Persons who are in a dependent or employment relationship with the auditor
3. For test persons: Exclusion, if they carry a known pain-relevant genetic variant/mutation or suffer from a chronic pain disorder analogous to migraine or chronic back pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: SFN Patients (Group A): Patients diagnosed with Small Fibre Neuropathia Healthy Volunteers (Group B): Healthy grown-up Volunteers Patients undergoing chemotherapy (Group C): Patients with imminent initiation of neurotoxic chemotherapy in cancer with solid tumors (preferably of the gastrointestinal tract) with the side-effect of SFN development. There are no plans for follow-up recruitment in case no neuropathy develops after chemo.
  Healthy Volunteers PREPs (Group D): Healthy grown-up Volunteers. Four subjects (2 male, 2 female) from each of the age decades 20-29, 30-39, 40-49, 50-59, 60-69.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
PainWatch Data | 12 months
  pulse rate (/min)
PainWatch Data | 12 months
  number of steps
PainWatch Data | 12 months
  pain perception via App (Questionnaire, pain scale 1-10)
Weather Data tracked according to GPS Location | 12 months
  Temperature (°C)
Weather Data tracked according to GPS Location | 12 months
  Air pressure (Pa)
Weather Data tracked according to GPS Location | 12 months
  Humidity (%)
Test result QST | 12 months
  Measurement exclusively above the back of the foot that is clinically more severely affected by the SFN, in a balanced row alternately above the right or left foot; one back of the foot as test site per subject
Test result PREP (over the same back of the foot as in QST measurement) | 12 months
  P1 Latency (ms)
Test result PREP (over the same back of the foot as in QST measurement) | 12 months
  Peak-to-Peak (microV)
Test result PREP (over the same back of the foot as in QST measurement) | 12 months
  Current intensity (mA)
Result SF 36 Questionnaire | 12months
  Result SF 36 Questionnaire (different scales per question)
Results of the Multi-Electrode Array investigations | 12 months
  Spontaneous activity
Results of the Multi-Electrode Array investigations | 12 months
  Synchronicity
Results of the Multi-Electrode Array investigations | 12 months
  Field potential properties
Results of the Multi-Electrode Array investigations | 12 months
  Activity inducing stimuli
Efficiency of reprogramming and differentiation of iPS cells | 12 months
  Success of differentiation will be measured by flow cytometry at around d10 of differentiation. The percentage of p75 (CD271)-expressing cells will be meassured. The differentiation is defined as successful if more than 30% of cells express p75. Only those differentiations will be used for MEA-Recordings.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Rolke, Prof. Dr., Principal Investigator — Universitätsklinikum Aachen, AöR
Locations (1):
- Uniklinik RWTH Aachen, Klinik für Palliativmedizin, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lacomis D. Small-fiber neuropathy. Muscle Nerve. 2002 Aug;26(2):173-88. doi: 10.1002/mus.10181. PMID 12210380
- [Background] Devigili G, Tugnoli V, Penza P, Camozzi F, Lombardi R, Melli G, Broglio L, Granieri E, Lauria G. The diagnostic criteria for small fibre neuropathy: from symptoms to neuropathology. Brain. 2008 Jul;131(Pt 7):1912-25. doi: 10.1093/brain/awn093. Epub 2008 Jun 4. PMID 18524793
- [Background] Rolke R, Rolke S, Hiddemann S, Mucke M, Cuhls H, Radbruch L, Elsner F, Peuckmann-Post V. [Update palliative pain therapy]. Internist (Berl). 2016 Oct;57(10):959-970. doi: 10.1007/s00108-016-0126-7. German. PMID 27631529
- [Background] Dworkin RH, O'Connor AB, Kent J, Mackey SC, Raja SN, Stacey BR, Levy RM, Backonja M, Baron R, Harke H, Loeser JD, Treede RD, Turk DC, Wells CD. Interventional management of neuropathic pain: NeuPSIG recommendations. Pain. 2013 Nov;154(11):2249-2261. doi: 10.1016/j.pain.2013.06.004. Epub 2013 Jun 6. PMID 23748119
- [Background] Coluzzi F, Rolke R, Mercadante S. Pain Management in Patients with Multiple Myeloma: An Update. Cancers (Basel). 2019 Dec 17;11(12):2037. doi: 10.3390/cancers11122037. PMID 31861097
- [Background] Meents JE, Bressan E, Sontag S, Foerster A, Hautvast P, Rosseler C, Hampl M, Schuler H, Goetzke R, Le TKC, Kleggetveit IP, Le Cann K, Kerth C, Rush AM, Rogers M, Kohl Z, Schmelz M, Wagner W, Jorum E, Namer B, Winner B, Zenke M, Lampert A. The role of Nav1.7 in human nociceptors: insights from human induced pluripotent stem cell-derived sensory neurons of erythromelalgia patients. Pain. 2019 Jun;160(6):1327-1341. doi: 10.1097/j.pain.0000000000001511. PMID 30720580
- [Background] Mucke M, Cuhls H, Radbruch L, Baron R, Maier C, Tolle T, Treede RD, Rolke R. [Quantitative sensory testing]. Schmerz. 2014 Dec;28(6):635-46; quiz 647-8. doi: 10.1007/s00482-014-1485-4. German. PMID 25403802
- [Background] Lefaucheur JP, Ahdab R, Ayache SS, Lefaucheur-Menard I, Rouie D, Tebbal D, Neves DO, Ciampi de Andrade D. Pain-related evoked potentials: a comparative study between electrical stimulation using a concentric planar electrode and laser stimulation using a CO2 laser. Neurophysiol Clin. 2012 Jun;42(4):199-206. doi: 10.1016/j.neucli.2011.12.003. Epub 2012 Jan 20. PMID 22632868
- [Background] Hansen N, Obermann M, Uceyler N, Zeller D, Mueller D, Yoon MS, Reiners K, Sommer C, Katsarava Z. [Clinical application of pain-related evoked potentials]. Schmerz. 2012 Feb;26(1):8-15. doi: 10.1007/s00482-011-1117-1. German. PMID 22134376
- [Background] Jenkinson C, Coulter A, Wright L. Short form 36 (SF36) health survey questionnaire: normative data for adults of working age. BMJ. 1993 May 29;306(6890):1437-40. doi: 10.1136/bmj.306.6890.1437. PMID 8518639
- [Background] Lee J, Mawla I, Kim J, Loggia ML, Ortiz A, Jung C, Chan ST, Gerber J, Schmithorst VJ, Edwards RR, Wasan AD, Berna C, Kong J, Kaptchuk TJ, Gollub RL, Rosen BR, Napadow V. Machine learning-based prediction of clinical pain using multimodal neuroimaging and autonomic metrics. Pain. 2019 Mar;160(3):550-560. doi: 10.1097/j.pain.0000000000001417. PMID 30540621